CLINICAL TRIAL: NCT01237002
Title: Safety of Intermittent Pringle Maneuver Cumulative Time Exceeding 120 Min in Liver Resection
Brief Title: Pringle Time Exceeding 120 Min in Liver Resection
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Guido Torzilli, MD, PhD, Liver Surgery Unit, Third Department of Surgery, University of Milan, IRCCS Istituto Clinico Humanitas
Other Study IDs: Pringle 120 minutes
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-10

CONDITIONS: Tolerance of the Liver
Keywords: Liver ischemia; Pringle time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: 117 patients with cumulative clamping time between 60 and 120 minutes
- Group 2: 72 patients with cumulative clamping time longer than 120 minutes

SUMMARY:
Intermittent Pringle's maneuver is widely used to limit blood loss during hepatectomy, without an established time-limit. However, many authors claims its danger for patients' outcome. The investigators check the short term outcome of a consecutive cohort of patients who underwent hepatectomy with intermittent clamping exceeding 120 minutes.

ELIGIBILITY:
Inclusion Criteria:

* patients in whom total cumulative clamping time exceeded 60 minutes.

Exclusion Criteria:

* patients in whom total cumulative clamping time was less than 60 minutes

Ages: 29 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among 426 consecutive patients who underwent hepatectomy, we retrospectively selected 189 patients with clamping time exceeded 60 minutes: 117 having intermittent Pringle maneuver less 120 minutes and 72 having clamping time exceeding 120 minutes were analysed.
Sampling Method: Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2005-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Torzilli, MD, PhD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- IRCCS Istituto Clinico Humanitas, Rozzano, Milan, Italy

REFERENCES:
- [Background] Belghiti J, Noun R, Malafosse R, Jagot P, Sauvanet A, Pierangeli F, Marty J, Farges O. Continuous versus intermittent portal triad clamping for liver resection: a controlled study. Ann Surg. 1999 Mar;229(3):369-75. doi: 10.1097/00000658-199903000-00010. PMID 10077049
- [Background] Elias D, Desruennes E, Lasser P. Prolonged intermittent clamping of the portal triad during hepatectomy. Br J Surg. 1991 Jan;78(1):42-4. doi: 10.1002/bjs.1800780115. PMID 1998862
- [Derived] Torzilli G, Procopio F, Donadon M, Del Fabbro D, Cimino M, Montorsi M. Safety of intermittent Pringle maneuver cumulative time exceeding 120 minutes in liver resection: a further step in favor of the "radical but conservative" policy. Ann Surg. 2012 Feb;255(2):270-80. doi: 10.1097/SLA.0b013e318232b375. PMID 21975322